CLINICAL TRIAL: NCT01477892
Title: Evaluation of Safety and Efficacy of Remifentanil in Preterm Infant
Brief Title: Evaluation of Safety and Efficacy of Remifentanil in Pediatric Population
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ajou University School of Medicine (Other); Severance Hospital (Other)
Responsible Party: Principal Investigator, Han-Suk Kim, Assist Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: RFTN-01; 11172_291 (Other: Korea Food and Drug Administrator)
Record Dates: First submitted 2011-11-10; First posted 2011-11-23 (Estimated); Results first posted 2013-09-13 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-09

CONDITIONS: Infant, Preterm
MeSH Terms: conditions — Premature Birth | interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low dose remifentanil (Experimental): continuous infusion of remifentanil 0.1mcg/kg/min
  Interventions: Drug: low dose remifentanil
- high dose remifentanil (Active Comparator): continuous infusion of remifentanil 0.25mcg/kg/min
  Interventions: Drug: low dose remifentanil

INTERVENTIONS:
Drug: low dose remifentanil — non-inferiority test for low dose remifentanil 0.1mcg/kg/min compared with high dose remifentanil 0.25mcg/kg/min in pain control
  Other Names: high dose remifentanil

SUMMARY:
The purpose of this study is to evaluate safety and efficacy of continuous infusion of remifentanil in preterm infant with mechanical ventilator for control of procedural pain using two different dosage of remifentanil.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants mechanically ventilated
* requiring peripherally induced central catheterization
* with informed consent of their parents

Exclusion Criteria:

* major congenital anomalies
* cardiopulmonary instability
* use of sedative, antiepileptic drugs or anesthetic drugs
* grade III or IV intraventricular hemorrhage

Max Age: 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2011-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Children's Hospital, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This noninferiority randomized, double-blind, controlled trial was conducted at the NICU of Seoul National University Children's Hospital and Ajou University Hospital between November 2011 and April 2012
Groups:
- High Dose Remifentanil: continuous infusion of remifentanil 0.25mcg/kg/min
  low dose remifentanil : non-inferiority test for low dose remifentanil 0.1mcg/kg/min compared with high dose remifentanil 0.25mcg/kg/min in pain control
- Low Dose Remifentanil: continuous infusion of remifentanil 0.1mcg/kg/min
  low dose remifentanil : non-inferiority test for low dose remifentanil 0.1mcg/kg/min compared with high dose remifentanil 0.25mcg/kg/min in pain control
Period: Overall Study
Arm/Group | High Dose Remifentanil | Low Dose Remifentanil
Started | 7 | 7
Completed | 7 | 5
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Remifentanil | Low Dose Remifentanil | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 5 | 12
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 7 | 5 | 12
Gestatonal age [Median (Full Range); unit: days] | 183 (0.03) [171 to 214] | 181 (0.03) [171 to 214] | 182 (0.03) [171 to 223]

OUTCOME MEASURES:

1. Primary Outcome: Premature Infant Pain Profile
Description: P0-P2 units on a scale
  ; changes in PIPP from baseline (P0) to procedure (needle puncture, P2)
  PIPP (preterm infant pain profile)
  * min 0 ~ max 21
  * higher pain scale on higher score
Time Frame: first puncture of skin(P0), 10min after remifentanil infusion (P1), 15min after remifentanil infusion (needle puncture, P2), 10min after remifentanil stop
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High Dose Remifentanil | Low Dose Remifentanil
Number analyzed (Participants) | 7 | 5
units on a scale | -0.60 (5.32) | 1.43 (3.10)

2. Secondary Outcome: Adverse Reaction
Description: bradycardia, hypotension, apnea, desaturation
Time Frame: during and after 10min of remifentanil continous infusion
Measure: Number; unit: participants
Arm/Group | High Dose Remifentanil | Low Dose Remifentanil
Number analyzed (Participants) | 7 | 5
participants
  Apnea | 3 | 0
  Bradycardia | 1 | 0
  Hypotension | 0 | 0

ADVERSE EVENTS:
Time Frame: during remifentanil infusion
Arm/Group | High Dose Remifentanil | Low Dose Remifentanil
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 3/7 | 0/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Remifentanil (N=7) | Low Dose Remifentanil (N=5)
apnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) — no self respiration for 20 sec
bradycardia (Cardiac disorders) | 1 (1) | 0 (0) — heart rate below 100/min

LIMITATIONS AND CAVEATS:
relatively small numbers of subjects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No